CLINICAL TRIAL: NCT07026253
Title: Comparative Analysis of Delirium in Older Patients Treated With Selected Antibiotics: a Prospective Cohort Study
Brief Title: Comparative Analysis of Delirium in Older Adults Treated With Ceftazidime, Cefepime, or Ceftriaxone
Acronym: CAD-CEF
Status: Recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0108470
Record Dates: First submitted 2025-04-28; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-08

CONDITIONS: Delirium
Keywords: cephalosporins; Antibiotics
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ceftazidime Group: A cohort of at least 40 older-adult patients (≥65 years) receiving ceftazidime for the treatment of various infections.
- Cefepime Group: A group of a minimum of 40 elderly patients treated with cefepime for confirmed or suspected infections.
- Ceftriaxone Group: This cohort will include at least 40 older adult inpatients receiving ceftriaxone as part of their anti-infective regimen

SUMMARY:
The goal of this observational study is to learn if the use of ceftazidime, cefepime, and ceftriaxone impacts the incidence of delirium in elderly patients (aged 65 and older) with infections. The main questions it aims to answer are:

Does the administration of these antibiotics increase the incidence of delirium in elderly patients? How do renal and hepatic dose adjustments affect the likelihood of delirium? Researchers will observe elderly patients receiving either ceftazidime, cefepime, or ceftriaxone for infection management to see if these antibiotics contribute to the onset of delirium, and then assessing the severity of the delirium.

Participants will:

Be assessed for delirium using the CAM (Confusion Assessment Method) at 2, 4, and 6 days after starting treatment.

Have their QSOFA (Quick Sequential Organ Failure Assessment) and NEWS (National Early Warning Score) tracked to evaluate their overall health status.

Undergo dose adjustments based on renal and hepatic function as part of their treatment.

Use the DRS.R89 score to assess delirium if it occurred.

DETAILED DESCRIPTION:
This observational study aims to assess the incidence, severity, and recovery of delirium in older adult patients treated with ceftazidime, cefepime, or ceftriaxone for infections. Delirium onset and severity will be monitored using the Confusion Assessment Method (CAM) and the Delirium Rating Scale (DRS-R98), alongside the Sequential Organ Failure Assessment (SOFA) scores, and National Early Warning Score (NEWS) for assessing the severity of infection. Key variables include the presence of delirium at Days 2, 4, and 6, and evaluating the severity of delirium and recovery time, as well as the impact of renal and hepatic dose adjustments. By examining these factors, the study seeks to provide insights into safer antibiotic use and dosing strategies in elderly patients, with the goal of reducing delirium risk and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Older adult patients aged 65 years or above.
* Hospitalized patients in Alexandria university hospitals diagnosed with infection and treated with selected cephalosporins (Ceftriaxone, Ceftazidime, or Cefepime).
* Patients without a history of Pre-existing delirium prior to hospitalization.

Exclusion Criteria:

* Patients with contraindications or allergies to cephalosporins.
* Patients with septic shock.
* Current use of medications known to cause delirium (anticholinergics, benzodiazepines, or opioid analgesics).
* Current or recent substance abuse (patients with a history of alcohol or drug abuse within the past year, or currently undergoing withdrawal). 5. Recent surgical procedures (patients who have undergone major surgery, particularly those requiring general anesthesia, within the last 30 days).
* Electrolyte imbalance (patients with severe electrolyte disturbances such as hypernatremia, hyponatremia, hypercalcemia or hypocalcemia at the time of study entry).
* Patients with End-stage renal disease requiring dialysis.
* Patients with severe liver disease (e.g., Child-C).
* Pain management issues: Patients with severe, uncontrolled pain that might independently affect cognitive function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients aged 65 or older at Alexandria University Hospitals receiving Ceftriaxone, Ceftazidime, or Cefepime.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium Diagnosed by Confusion Assessment Method (CAM) | Within 6 days after initiation of antibiotic treatment
  : Determine the incidence of delirium in older-adult patients treated with selected cephalosporins, diagnosed using the Confusion Assessment Method (CAM).
  Units of Measure: Number of participants with CAM-positive delirium Details: The CAM is a validated diagnostic tool for delirium based on four features: (1) acute onset and fluctuating course, (2) inattention, (3) disorganized thinking, and (4) altered level of consciousness. Delirium is diagnosed when both features 1 and 2 are present, and either feature 3 or 4.
  Incidence will be calculated as the number of patients who meet the CAM criteria divided by the total number of patients in each treatment arm.

SECONDARY OUTCOMES:
Delirium severity | On the day of delirium diagnosis
  Description: Severity of delirium measured using the Delirium Rating Scale-Revised-98 (DRS-R-98).
  Units of Measure: DRS-R-98 score (0-39 for severity scale) Delirium Rating Scale-Revised-98 (DRS-R-98) is a standardized tool used to assess the severity and presence of delirium. It includes 16 items - 13 severity items and 3 diagnostic items - and is rated based on clinical observation and patient interaction.
  Scoring Overview:
  13 severity items are scored from 0 to 3 (maximum score = 39) 3 diagnostic items are scored from 0 to 3 (maximum score = 9) Total maximum score = 46
Length of hospital stay | From hospital admission until discharge, assessed up to 90 days.
  Total number of days the patient remained hospitalized during the study period.
Mortality rate | From hospital admission until in-hospital death or discharge, assessed up to 90 days
  Proportion of patients who died during hospitalization period.
Time to delirium onset | From the date of antibiotic initiation until the first documented CAM-positive delirium event, assessed up to 6 days
  Number of days from the initiation of the antibiotic to the onset of clinically confirmed delirium (via Confusion Assessment Method [CAM]).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospitals, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No